CLINICAL TRIAL: NCT02125305
Title: A Phase I Clinical Study to Investigate the Pharmacokinetics and Pharmacodynamics of Metformin in Elderly Healthy Male Volunteers
Brief Title: Clinical Study to Investigate the Pharmacokinetics and Pharmacodynamics of Metformin in the Elderly
Acronym: ME01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae Yong Chung, M.D., Ph.D, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ME01
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Healthy Elderly
Keywords: Metformin; Pharmacokinetics/ Pharmacodynamics
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin (Experimental): Metformin 750mg(D1), Metformin 500mg(D2)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin
  Other Names: Diabex

SUMMARY:
This study aims to investigate the pharmacokinetics/pharmacodynamics metformin IR after oral administration in healthy elderly male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 65-85 years with a body mass index (BMI) of 18-28 kg/m2
* Good health based on complete medical history, physical examinations, vital signs, electrocardiography (ECG), and clinical laboratory evaluations including hematology (blood cell count, hemoglobin, and platelet count), liver function test (aspartate aminotransferase (AST), alanine aminotransferase (ALT), and bilirubin), serum creatinine, blood glucose and urinalysis

Exclusion Criteria:

* If they had clinically relevant disorders
* Past history of diabetes or clinical findings to suspect diabetes
* Abnormal clinical laboratory values (i.e., platelets ≤ 75,000/mm3, hemoglobin ≤ 9 g/dL, neutrophils absolute ≤ 1000/mm3, fasting glucose > 126mg/dL, creatinine ≥ 1.5 mg/dL, or AST, ALT > 3 × upper limit of normal)

Ages: 65 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-08; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
AUC(area under the plasma concentration-time curve) | Predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12h postdose
  AUC(area under the plasma concentration-time curve), Cmax(maximum plasma concentration), t1/2

SECONDARY OUTCOMES:
AUGC(total area under the serum concentration-time curve for glucose concentration) | predose and 15, 30, 45, 60, 90, 120 min oral glucose tolerance test
  AUG (total area under the serum concentration-time curve for glucose) Gmax(maximum serum glucose concentration)

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Yong Chung, M.D., Ph.D., Principal Investigator — Department of Clinical Pharmacology and Therapeutics, Seoul National University Bundang hospital
Locations (1):
- Seoul National University Bundang Hospital, Seoul, South Korea